CLINICAL TRIAL: NCT07056699
Title: Protocol V: San Antonio Site Sub Study: Can Pioglitazone Block SGLT2 Inhibitor-induced Stimulation of Lipolysis, Ketone Production and Liver Glucose Production in Type I Diabetic Patients
Brief Title: SGLT2i, Pioglitazone, and Ketone Production in T1D
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: The University of Texas Health Science Center at San Antonio (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: STUDY00001633 - 504078; R01DK024092 (NIH)
Record Dates: First submitted 2025-06-26; First posted 2025-07-09 (Actual); Last update posted 2025-11-10 (Actual); Status verified 2025-11

CONDITIONS: Type1diabetes
Keywords: Selective Glucose Cotransporter 2 inhibitors (SGLT2i); Dapagliflozin; Pioglitazone
MeSH Terms: interventions — dapagliflozin; Pioglitazone

STUDY DESIGN:
Intervention Model Description: A cluster randomized, double-blind, placebo-controlled mechanistic study
Who Masked: Participant, Investigator
Masking Description: At week 16, subjects will be randomized to receive in a double-blinded fashion pioglitazone or placebo for 16 weeks.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Experimental study drug for T1D (Experimental): Dapagliflozin (10 mg/day) + Pioglitazone (15 mg/day for 2 weeks, then 30 mg/day for 14 weeks)
  Interventions: Drug: Dapagliflozin 10mg Tab; Drug: Pioglitazone 15 MG and 30mg
- Placebo Group for T1D (Placebo Comparator): Dapagliflozin (10 mg/day) + Placebo (for 16 weeks)
  Interventions: Drug: Dapagliflozin 10mg Tab; Other: Placebo

INTERVENTIONS:
Drug: Dapagliflozin 10mg Tab — Dapagliflozin (10 mg/day)
  Other Names: Farxiga
Drug: Pioglitazone 15 MG and 30mg — Pioglitazone (15 mg/day for 2 weeks, then 30 mg/day for 14 weeks)
  Other Names: Actos
  Arms: Experimental study drug for T1D
Other: Placebo — Inert placebo for Pioglitazone
  Other Names: Inert substance
  Arms: Placebo Group for T1D

SUMMARY:
Participants are being asked to be in a research study. Scientists do research to answer important questions which might help change or improve treatment of participants disease in the future.

In patients with Type 1 Diabetes (T1D), Dapagliflozin a Selective Glucose Transporter 2 Inhibitor (SGLT2i) is known to increase production of glucose in the liver, increase breakdown of fats (lipolysis), and increase production of ketones (ketogenesis). Ketones are chemicals produced by the liver when the body breaks down fat for energy instead of glucose. When the level of ketones in the body becomes too high, a condition called ketoacidosis develops. In this study, the study team will investigate whether adding pioglitazone (a medication commonly used to treat type 2 diabetes), can reduce the Dapagliflozin - induced liver glucose production, fat break down (lipolysis) and ketone body production (ketogenesis) in patients with Type 1 Diabetes (T1D).

DETAILED DESCRIPTION:
The purpose of this research study is to investigate the effects of Dapagliflozin and Pioglitazone in the body - specifically, on liver glucose production, breakdown of fat, and ketone production in Type 1 Diabetic patients treated with insulin. Subjects with type 1 diabetes mellitus (T1DM) can't make insulin because their pancreas doesn't work properly. This means they need insulin injections to control their blood sugar. But using insulin can sometimes cause low blood sugar and weight gain, making it harder for insulin to work and requiring higher doses. Finding other medicines that can help lower blood sugar in people with T1DM and can be used along with insulin would make it easier to manage their blood sugar.

Dapagliflozin is in a class of drugs known as Selective Glucose Cotransporter 2 inhibitors (SGLT2i) and has been shown to effectively lower blood sugar concentration in type 1 diabetes mellitus (T1DM) patients. These drugs lower blood glucose levels by preventing or reducing the re-absorption of glucose in the kidneys. This results in the release of glucose into the urine. At the same time, Selective Glucose Transporter 2 Inhibitor (SGLT2i) drugs stimulate glucose production by the liver, which helps compensate for the loss of glucose into the urine. Also, the use of dapagliflozin in patients with type 1 diabetes was associated with increased risk of ketoacidosis. Ketoacidosis is a serious condition that occurs when the body produces high levels of ketones, leading to increased acidity in the blood. Pioglitazone is in a class of thiazolidinediones and is commonly used to treat high blood sugar levels caused by type 2 diabetes. The investigators believe that the addition of pioglitazone, to dapagliflozin will prevent the risk of ketoacidosis associated with dapagliflozin, and will cause a large reduction in plasma glucose concentration in type 1 diabetes (T1DM) patients.

ELIGIBILITY:
Inclusion Criteria:

1. Age >18 years
2. T1DM
3. Other than diabetes, subjects must be in good general health as determined by physical exam, medical history, Chem 20, CBC, TSH, urinalysis, and EKG.
4. Fasting C-peptide concentration <0.7 ng/ml
5. Poor glycemic control (HbA1c=7.0-11.0%)
6. Treatment with multiple daily insulin injections (basal plus prandial) or insulin pump
7. Total daily insulin dose ≥0.6 U/kg per day
8. Stable insulin dose (±4 units) in the preceding three months.
9. eGFR≥60 ml/min
10. Weight stable over the preceding 3 months (± 3 pounds) and who do not participate in an excessively heavy exercise program

Exclusion Criteria:

1. T2DM
2. Daily insulin dose <0.6 U/kg per day
3. Fasting C-peptide >0.7 ng/ml
4. HbA1c <7.0% or >11.0%
5. eGFR<60 ml/min
6. Hematuria in urine analysis
7. Pregnancy, lactating, positive pregnancy test or planning to become pregnant in the following year. Women of child-bearing potential will be requested to use at least two barrier methods before being enrolled in the study.
8. Major organ system disease which includes: (i) malignancy or history of malignancy including bladder cancer; (ii) Congestive heart failure or history of coronary heart disease or any other cardiac disease; (iii) chronic liver disease or LFT >3 times the upper normal level; (iv) History of alcohol or drug abuse; (v) History of chronic lung disease (e.g., COPD, asthma); (vi) history of rheumatic disease; (vii) History of chronic pancreatitis or pancreatic surgery; (viii) History of CVA or TIA (ix) Planned surgery during the study; (x) history of HIV infection or other immune compromised disease; and history of organ transplantation; (xi) patients who take medications, other than insulin, known to affect glucose metabolism, e.g., prednisone.
9. Evidence of proliferative diabetic retinopathy
10. Patients enrolled in a heavy exercise program
11. Patients on ketogenic diet
12. History of hospitalization for DKA, hypoglycemia or uncontrolled hyperglycemia in the preceding 6 month.
13. Presence of symptoms of poor glycemic control, e.g. polydipsia or polyurea
14. History of hypersensitivity to dapagliflozin or pioglitazone

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2026-01-30 (Estimated); Primary Completion 2027-06-01 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
Change in endogenous glucose production (EGP) | Baseline (Week 0) to Week 16
  Infusions of a tracer, ³H-glucose, will begin and continue until the end of the study.
  A single dose of empagliflozin (25 mg) by mouth will be taken at 900am. Blood samples will be collected minutes to assess how your body responds to the infused tracers.
  This tracer help to measure the rate of endogenous (liver) glucose production. The difference in levels of EGP will be reported from the beginning of the study to a second level taken 16 weeks later.
Change in ketone body production ( ketogenesis) | Baseline (Week 0) to Week 16
  Infusions of tracers, ³H-glucose and U-2H-glycerol or 14C-Glycerol, will begin and continue until the end of the study.
  A single dose of empagliflozin (25 mg) by mouth will be taken at 900am. Blood samples will be collected to assess how your body responds to the infused tracers.
  This tracer help to measure the rate of ketone body production (ketogenesis). The difference in levels of ketones will be reported from the beginning of the study to a second level taken 16 weeks later.
Change in lipolysis (fat breakdown) | Baseline (Week 0) to Week 16
  Infusions of tracers, U-H-14C-Glycerol or 2H-Glycerol, will begin and continue until the end of the study.
  A single dose of empagliflozin (25 mg) by mouth will be taken at 900am. Blood samples will be collected to assess how your body responds to the infused tracers.
  This tracer help to measure the rate of lipolysis (fat breakdown). The difference in levels of lipolysis will be reported from the beginning of the study to a second level taken 16 weeks later.

SECONDARY OUTCOMES:
Change in HbA1c from baseline (Week 0) to Week 16 | Baseline (Week 0) to Week 16
  HbA1c and CGM metrics provide clinically relevant data on glycemic control and variability. This endpoint assess the metabolic efficacy of adding pioglitazone to dapagliflozin in T1DM.
Change in plasma Free Fatty Acid (FFA) from baseline (Week 0) to Week 16. | Baseline (Week 0) to Week 16
  Measuring free fatty acids directly tests the hypothesis that pioglitazone reduces the risk of SGLT2 inhibitor-associated diabetic ketoacidosis (DKA) by suppressing FFA release.
Change in glycerol from baseline (Week 0) to week 16. | Baseline (Week 0) to Week 16
  To examine the effects of adding pioglitazone (15/30 mg/day) to dapagliflozin (10 mg/day) compared to dapagliflozin (10mg/day) plus placebo in T1DM patients, focusing on lipolysis changes over a 16-week treatment period.

CONTACTS AND LOCATIONS:
Overall Officials: Muhammad Abdul-Ghani, MD, Principal Investigator — The University of Texas Health Science Center at San Antonio; Ralph DeFronzo, MD, Principal Investigator — The University of Texas Health Science Center at San Antonio
Locations (1):
- Texas Diabetes Institute, San Antonio, Texas, United States

IPD SHARING:
Plan to Share IPD: Yes
Study participant research data, which is for purposes of statistical analysis and scientific reporting, will be transmitted to and stored at the Diabetes division at UT Health. This will not include the participant's contact or identifying information. Rather, individual participants and their research data will be identified by a unique study identification number. The study data entry and study management systems used by clinical sites and by Diabetes division at UT Health research staff will be secured, and password protected. At the end of the study, all study databases will be de-identified and archived at the Diabetes division at UT Health.
Supporting Information: Study Protocol, SAP
Time Frame: At the end of the study, after data analysis is complete.